CLINICAL TRIAL: NCT05447572
Title: FIT Combining FC for Predicting MH and Histology Remission in UC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Professor, Shandong University
Other Study IDs: 2022SDU-QILU-1
Record Dates: First submitted 2022-01-05; First posted 2022-07-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Ulcerative Colitis; Histology Remission; Fecal Calprotetin; FIT; Mucosal Healing
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Each colonoscopies will get common biospies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FIT combingning FC with colonscopy
  Interventions: Other: FIT + FC

INTERVENTIONS:
Other: FIT + FC — FIT + FC

SUMMARY:
Investigaters will perform a clinical trial to asess the abilitiy of qFIT and FC on predicting UC MH and histology remission.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis patients.

Exclusion Criteria:

* GI bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ulcerative colitis patients.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic value of FIT and/without FC on predicting MH | 2 weeks
  diagnostic value of FIT and/without FC on predicting MH, Mayo score will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided